CLINICAL TRIAL: NCT01883050
Title: Application for Self-Monitoring of Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas G. Allison, Ph.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-004546
Record Dates: First submitted 2013-06-04; First posted 2013-06-21 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Coronary Disease
Keywords: Coronary artery disease; Percutaneous Intervention; Stent; Balloon angioplasty; Angiogram; Coronary angiogram
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Monitoring of Software Application (Other): log into self monitoring software application from a home computer. Log on 3-4 times weekly for 12 weeks for important reminders, care tips and educational materials.
  Interventions: Device: Self Monitoring Software Application
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Device: Self Monitoring Software Application — Computer Software application to track health progress after interventional surgery
  Arms: Self Monitoring of Software Application

SUMMARY:
Patients who recently suffered a heart attack will use a smart-phone/computer application during cardiac rehabilitation to reduce their risk of a future attack, their re-hospitalizations, their cost of care, and increase their quality of life.

DETAILED DESCRIPTION:
The study will consist of two phases - an initial feasibility trial (Phase 1), followed by a randomized clinical trial (Phase 2). Once the Phase 1 trial is evaluated, Phase 2 will be implemented.

Phase 1 will consist of up to 35 participants to ensure that the software application is user-friendly, properly stores pertinent data, and has no technical glitches. All participants in Phase 1 will have access to the software application and will be asked to complete online questionnaires, at baseline and post cardiac rehab, to assess their quality of life and also their satisfaction with their care and the software application itself.

Phase 2 will consist of 65 participants. These participants will be randomized to either 1) Cardiac Rehab (CR) alone along with answering questionnaires regarding quality of life and satisfaction of care or 2) CR along with the software application and the quality of life, satisfaction of care and software application questionnaires. All participants (both Phase 1 and Phase 2) enrolled into the study will be status-post percutaneous coronary intervention (PCI). The potential participants will be asked to participate while still in the hospital and will be approached as soon as possible after agreeing to participate in CR,. The participants who enroll in Phase 2 will be randomized prior to discharge from the hospital.

All participants in Phase 1 and those in Phase 2 who randomize to the software application will be instructed on the use of either the desktop or smart-phone version of the software application. Baseline information, including participant name, date of birth, email address, and phone number, will be gathered from the participant at that time, and all characteristics will be entered by the participant and study coordinator into their own account in the application.

The study will follow all Phase 1 participants and those in Phase 2 who randomize to the software application for three months after hospital dismissal and evaluate the following:

* Weight/BMI, blood pressure, and heart rate
* Usual lab values already gathered for the participant such as lipids, Complete Blood Count (CBC), and HgbA1C
* Quality of life, disposition, and mood
* Participant compliance, satisfaction, and adherence to the application
* Re-hospitalizations, participants phone calls, and cost of care

During the second week of their CR an additional 30-60 minute educational session will be required so that the study coordinator can instruct the participant on the software application and how to use it.

We will also ask that participants "log in" to their online account at least 3-4 times weekly for important reminders, care tips, and educational materials. This will last the duration of their cardiac rehabilitation program (approximately 12 weeks). Specific examples of sections within the software application will pertain to medication adherence, diet, exercise, educational materials, and reviews of your medical profile.

Finally, we would ask that participants (all of Phase 1 and those who randomize to the software application in Phase 2) to complete online questionnaires, at baseline and post cardiac rehab. that assess their quality of life and also their satisfaction with their care and the software application itself. This will be used for both data purposes as well as in future improvements to the program. These individual surveys will take approximately 5 minutes to complete. Phase 2 study participants who do not randomize to the software application will be sent the quality of life and satisfaction of care questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Recently underwent PCI.
* Are eligible for enrollment to the Cardiovascular Health Clinic (CVHC)
* Do not have any physical impediments to physical activity
* Do not have any impediments to physically attending the Mayo Clinic's CVHC
* They are willing to incorporate the software application into their CR
* They must have access to the internet

Exclusion Criteria:

* - They are unable or unwilling to enroll in CR
* They are unable to physically attend Mayo Clinic's CVHC CR Program
* They are unwilling to incorporate the Personal Health Assistant into their CR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who completed all tasks in the application. | Baseline to 3 months
  These data will provide the best summary of usability of the application.

SECONDARY OUTCOMES:
User-reported satisfaction with application. | Baseline to 3 months
  These data will provide additional insights into how users view the application interface and help us modify the design to enhance compliance.

OTHER OUTCOMES:
Body weight | Baseline to 3 months
  Weight will be the most sensitive indicator that completion of the tasks assigned in the application lead to subsequent behavioral chance and reduction of cardiovascular risk.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Allsion, PHD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Widmer RJ, Senecal C, Allison TG, Lopez-Jimenez F, Lerman LO, Lerman A. Dose-Response Effect of a Digital Health Intervention During Cardiac Rehabilitation: Subanalysis of Randomized Controlled Trial. J Med Internet Res. 2020 Feb 26;22(2):e13055. doi: 10.2196/13055. PMID 32130116
- [Derived] Widmer RJ, Allison TG, Lennon R, Lopez-Jimenez F, Lerman LO, Lerman A. Digital health intervention during cardiac rehabilitation: A randomized controlled trial. Am Heart J. 2017 Jun;188:65-72. doi: 10.1016/j.ahj.2017.02.016. Epub 2017 Feb 20. PMID 28577682